CLINICAL TRIAL: NCT05065580
Title: Osteopathic Manipulative Treatment as an Adjunctive Treatment in Major Depressive Disorder
Brief Title: OMT as an Adjunctive Treatment in MDD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corewell Health South (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EGME#05-2021
Record Dates: First submitted 2021-09-23; First posted 2021-10-04 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Somatic Symptom Score (Active Comparator): Patients meeting PHQ-9 (Patient health Questionnaire)-9 with score greater than 10 with Somatic Symptom Score less than 7.
  These patients will receive the OMT treatment protocol and PHQ-9 and SSS scales will be recorded at 0, 4, and 8 weeks.
  Interventions: Procedure: Osteopathic Manipulative Treatment
- High Somatic Symptom Score (Active Comparator): Patients meeting PHQ-9 (Patient health Questionnaire)-9 with score greater than 10 with Somatic Symptom Score 8 or greater These patients will receive the OMT treatment protocol and PHQ-9 and SSS scales will be recorded at 0, 4, and 8 weeks.
  Interventions: Procedure: Osteopathic Manipulative Treatment

INTERVENTIONS:
Procedure: Osteopathic Manipulative Treatment — Individuals will receive the following techniques during weekly OMT (osteopathic manipulative techniques) for a duration of 8 weeks: 1. Suboccipital release 2. Vault hold. 3. Soft tissue techniques at the cervical and shoulder region 4.There will be NO high velocity low amplitude (HVLA) techniques

SUMMARY:
participants will be receiving OMT 1x/week for 8 weeks. Each appointment with be a duration of 30 minutes. Patients will be required to fill out PHQ-9 and SSS-8 questionnaires before beginning the study and following the conclusion of the study.

DETAILED DESCRIPTION:
Individuals will receive weekly OMT for a duration of 8 weeks. Primary assessment will be performed on initial visit, making note of the most severe somatic restrictions, but highest priority will be given to cervical and shoulder regions (most tension is noted here in patients with MDD). Focusing on only the cranial, cervical, and shoulder regions will allow for a more standardized approach to treatment.

Osteopathic manipulative treatment (OMT) is the manipulation of tissues (muscles, joints, fascia, etc.) that is used to help restore movement and function throughout the body by a combination of stretching, gentle pressure, and resistance. The techniques we have chosen to use will focus primarily on muscle and fascia in the cranial, cervical, and shoulder regions.

Cranial techniques used include:

Suboccipital release - this helps to relieve muscle and fascial tension surrounding the head and neck, patient is supine, physician places finger pads below occipital protuberance at the base of the occiput as patient's relaxes head and lets it rest on physician's finger pads, position is held until softening of musculature is felt

Vault hold - helps to restore cranial motion, patient is supine, physician places index finger on greater wing of sphenoid, middle finger on squamous portion of temporal bone, ring finger on mastoid process of temporal bone, and pinky finger on squamous portion of occipital bone, hands remain in this position to monitor cranial motion and determine if there is a dysfunction

They will NOT be performing any high velocity low amplitude (HVLA) techniques, which requires a rapid, therapeutic force within the motion of the joint (this is the technique that is often responsible for the "cracking" or "popping")

ELIGIBILITY:
Inclusion Criteria:

* patients 18-65, patients with diagnosis of MDD, PHQ-9 score > 10 at screening and baseline

Exclusion Criteria:

* history of mania, hypomania, or psychosis as defined in DSM V
* current substance abuse, including abuse within the previous 6 months
* patients with a cognitive disorder or dementia
* patients with other axis I diagnosis (anxiety disorders, dissociative disorders, etc.) that was primary in the past 6 months
* receiving other forms of manual therapy during study
* authors belief that there was significant suicidal risk
* changes in medication or psychotherapy within 6 weeks of starting study or during study period
* history of migraines
* presence of any other significant organic disease (infectious, cardiac, pulmonary, gastrointestinal, renal, etc.)
* other absolute contraindications to OMT (malignancy, infection, myelopathy, severe osteoporosis, increased ICP, intracranial bleeding, fractures, etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

PRIMARY OUTCOMES:
PHQ-9 (Patient Health Questionnaire) results post treatment | 8 weeks
  compare PHQ-9 results in the two groups based on SSS-8 (Somatic Symptom Score) score before and after treatment. PHQ-9 is a depression score ranging from 0 through 27. No depression 0-4, mild 5-9, moderate 10-14, moderately severe 15-19, severe 20-27. The SSS-8 ranges from 0 through 32. No to minimal symptoms range from 0 through 3, low from 4-7, medium 8-11\, high 12-15, very high 16-32.

CONTACTS AND LOCATIONS:
Locations (1):
- Lakeland Regional Healthcare, Saint Joseph, Michigan, United States

IPD SHARING:
Plan to Share IPD: No